CLINICAL TRIAL: NCT04642300
Title: Effect of Holmich Protocol and Myofascial Release Technique on Groin Pain in Tennis Players
Brief Title: Holmich Protocol and Myofascial Release Technique Effect on Groin Pain in Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00722 Rohail Babar
Record Dates: First submitted 2020-05-29; First posted 2020-11-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Sports Physical Therapy
Keywords: Groin pain; Holimch protocol; Myofascial release technique
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holmich Protocol (Active Comparator): Treatment will be administered three times a week (on even or odd days). The duration of each session was about 90 min for module 1 (first two weeks) and 120 min for module 2 (from the third week). From the third week, the athletes were asked to perform exercises from module 1 every other day, between the treatment sessions
  Interventions: Procedure: Holmich Protocol
- Myofascial Release Technique (Active Comparator): Treatment wiil be given twice a week as individual treatment by the physiotherapist. The duration of treatment is about 30 min.
  Interventions: Procedure: Myofascial Release Technique

INTERVENTIONS:
Procedure: Holmich Protocol — Module 1 (1st two weeks):
  i)Isometric adduction ii)Abdominal sit-ups iii)Isometric adduction iv)Compound abdominal sit-ups and hip flexion v)Balance exercise on wobble board vi)One-foot exercise on sliding board
  Module 2 (from 3rd week):
  i)Leg abduction and adduction exercise carried out in side lying ii)Low back extension exercise prone on the end of bench iii)One leg weight pulling abduction/adduction standing iv)Abdominal sit ups v)One leg coordination exercise vi)Training in sideways motion vii)Balance exercise on wobble board
  Arms: Holmich Protocol
Procedure: Myofascial Release Technique — 1. Transverse friction massage: 10 mins on painful area of adductor-tendon insertion into pubic bone
  2. Stretching of adductor muscles, hamstrings muscles and hip flexors:3 times and each stretch is 30s with Contract relax technique
  Arms: Myofascial Release Technique

SUMMARY:
The aim of this study is to determine the effect of Homlich Protocol and Myofacial release technique on groin pain in tennis players. A total of 14 players will be included in the clinical trail. There will be one group of 7 players in which Holmich protocol will be applied while in the other group of 7 players will be given Myofascial Release Technique which includes Transverse friction massage and Stretching. Data will be collected by outcome measures before and after the exercise protocol is given. Treatment will be administered three times a week (on even or odd days). The duration of Holmich Protocol each session is about 90 min for module 1 (first two weeks) and 120 min for module 2 (from the third week). From the third week, the athletes will be asked to perform exercises from module 1 every other day, between the treatment sessions. While passive treatment will be given for 30 mins per session. During the treatment course and before the final evaluation, no athletic activity will be permitted . Injuries data will be collected prospectively by respective coaches. Coaches will be trained for identification and classification of injuries.

DETAILED DESCRIPTION:
Groin pain arising from sports injuries is widespread, especially among those who participate in sports that involve repetitive rotational movements such as kicking and turning as in soccer. This type of injury is the fourth most common sports injury, with soccer players suffering from long-term symptoms and frequent relapses. The injury rate is 1.015-1.133 per 1000 hours of play, which is equivalent to 11%-16% of all sports injuries. The prognosis for exercise- related groin pain is not clear. Injured athletes may be forced to wait a long time before returning to sports activity free of restriction.

It is known that adductor-related groin injuries are the most common cause of groin injury, accounting for 69% of groin injuries in football and 58% across all forms of sport. As limited range of hip abduction and hip internal rotation and decreased hip adductor strength (absolute and comparative to the hip abductors) are considered potential risk factors for groin injury. Adductor-related groin pain is often treated without surgery. Among different conservative approaches, it appears that exercise therapy (ET) is more effective than other conservative treatment methods such as electrotherapy, manual therapy or steroid injections. Unfortunately, however, many important factors including frequency, duration and the exact amount of resistance or perceived exertion to be used in the ET protocols have not been carefully recorded in clinical trials. To our best knowledge, the randomised clinical trial carried out by Holmich et al in 1999 still offers the best evidence for the effectiveness of exercise as a prescription for the treatment of adductor-related groin pain. Holmich et al collated the results of ET (based on isometric and isotonic strengthening of the hip abductor/adductor and the abdominal muscles) with results from physiotherapy. They evaluated successful treatment (based on pain measures), patients' subjective global assessments and their return to sport without groin pain at the same level as before the injury. 'Successful treatment' as described in their study is an unfeasible and non-validated measure for evaluating outcome; on the other hand, the published results by Holmich et al was not compared with any such other treatment.

Yousefzadeh A et al conducted a study which checked the effect of Holmich Protocol on groin pain and its results showed to be an effective treatment.

Weir A et al performed multi modal treatment(MMT) in comparison to exercise therapy(ET), results showed MMT to be more effective then ET.

Sernar A et al did a systemic review on treatment of groin players which showed low quality studies present for groin injury management.

Holmich P et al performed a randomized trial on effects of active physical training(AT) on groin pain, results showed AT to be very effective on groin pain.

Kalichman L and Ben David C did a narrative review on the effect of self-myofascial release(SMFR) and concluded that there was a significant increase in joint range of motion and no decrease in muscle force.

Timothy C.Mauntel et al performed myofascial release technique to increase physical performance measurements to check its effectiveness. The systematic review observed a significant change in range of motion but no significant change in muscle function.

Melih Paksoy and Umit Sekmen performed a review of current diagnosis and treatment modilities which showed that response rates to conservative treatment for inguinal pain is very low.

Dines et al performed a study on tennis injuries and showed that groin pain to be present around 3% to 21%.

In the current study, we will reproduce Holmich et al research along with Myofascial release technique to treat long-standing adductor-related groin pain (LSAGP) and analyse the short-term flow of alterations in pain and functional ability. Furthermore, as limited range of hip abduction and hip internal rotation and decreased hip adductor strength (absolute and comparative to the hip abductors) are considered potential risk factors for groin injury, we will also measure these variables as our outcomes. The purpose of this study is to obtain an objective evaluation of the effect of Holmich protocol and Myofascial release technique to compare which is better in treating LSAGP.

ELIGIBILITY:
Inclusion Criteria:

* Male Gender
* Age: 18 - 35 years
* Groin pain for at least 2 months
* 3 - 7 pain score on NPRS
* Playing Sports for atleast 1 year

Exclusion Criteria:

* Femoral or inguinal hernia
* Chronic urinary tract disorder or prostatitis
* Disease, fracture of the pelvis or the lower limbs inhibiting the participant from the completing the treatment plan
* Entrapment of the genitofemoral or back pain felt between T10 and L5 levels and consisting of the facet joints
* Virulent Ilioinguinal nerve
* Inability to follow the active physical training plan
* Use of non-steroidal anti-inflammatory drugs during the study
* Participation in principled strength training of the hip adductors for more than once a week in the 6 months prior to the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Hip Range of motion | 8 Weeks
  The hip range of motion including abduction, adduction, external and internal rotation in 90°of flexion will be measured by an adjustable goniometer.
T-Agility TEST | 8 Weeks
  Set out four cones 5 yards = 4.57 m, 10 yards = 9.14 m. The subject starts at cone A. On the command of the timer, the subject sprints to cone B and touches the base of the cone with their right hand. They then turn left and shuffle sideways to cone C, and also touches its base, this time with their left hand. Then shuffling sideways to the right to cone D and touching the base with the right hand. They then shuffle back to cone B touching with the left hand, and run backwards to cone A. The stopwatch is stopped as they pass cone A
Edgren Side Test (ESST) | 8 Weeks
  Five cones or lines are placed in a line, three feet apart (12 feet total between the two outside cones). The starting position is at the centre cone, facing forward with feet straddling the center line. At the command 'go', the participant sidesteps to the right until their right foot touches or crosses the outside cone or tape mark. The participant then sidesteps to the left until their left foot touches or crosses the left outside cone or tape mark. The participant sidesteps back and forth to the outside cones as rapidly as possible for 10 seconds.
Triple Hop Test (THT) | 8 Weeks
  In the triple hop test, the aim is to jump as far as possible on a single leg three consecutive times, without losing balance and landing firmly. The distance is measured from the start line to the heel of the landing leg. The goal is to have a less than 10% difference in hop distance between the injured limb and uninjured limb.
Visual Analogue Scale Pain Score (VAS) | 8 Weeks
  The visual analog scale (VAS) scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm). The values can be used to track pain progression for a patient or to compare pain between patients with similar conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faheem Afzal, *PhD, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caudill P, Nyland J, Smith C, Yerasimides J, Lach J. Sports hernias: a systematic literature review. Br J Sports Med. 2008 Dec;42(12):954-64. doi: 10.1136/bjsm.2008.047373. Epub 2008 Jul 4. PMID 18603584
- [Background] Hawkins RD, Hulse MA, Wilkinson C, Hodson A, Gibson M. The association football medical research programme: an audit of injuries in professional football. Br J Sports Med. 2001 Feb;35(1):43-7. doi: 10.1136/bjsm.35.1.43. PMID 11157461
- [Background] Walden M, Hagglund M, Werner J, Ekstrand J. The epidemiology of anterior cruciate ligament injury in football (soccer): a review of the literature from a gender-related perspective. Knee Surg Sports Traumatol Arthrosc. 2011 Jan;19(1):3-10. doi: 10.1007/s00167-010-1172-7. Epub 2010 Jun 9. PMID 20532868
- [Background] Holmich P, Thorborg K, Dehlendorff C, Krogsgaard K, Gluud C. Incidence and clinical presentation of groin injuries in sub-elite male soccer. Br J Sports Med. 2014 Aug;48(16):1245-50. doi: 10.1136/bjsports-2013-092627. Epub 2013 Aug 16. PMID 23956334
- [Background] Weir A, Jansen JA, van de Port IG, Van de Sande HB, Tol JL, Backx FJ. Manual or exercise therapy for long-standing adductor-related groin pain: a randomised controlled clinical trial. Man Ther. 2011 Apr;16(2):148-54. doi: 10.1016/j.math.2010.09.001. Epub 2010 Oct 16. PMID 20952244
- [Background] Almeida MO, Silva BN, Andriolo RB, Atallah AN, Peccin MS. Conservative interventions for treating exercise-related musculotendinous, ligamentous and osseous groin pain. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD009565. doi: 10.1002/14651858.CD009565.pub2. PMID 23740671
- [Background] Holmich P, Uhrskou P, Ulnits L, Kanstrup IL, Nielsen MB, Bjerg AM, Krogsgaard K. Effectiveness of active physical training as treatment for long-standing adductor-related groin pain in athletes: randomised trial. Lancet. 1999 Feb 6;353(9151):439-43. doi: 10.1016/S0140-6736(98)03340-6. PMID 9989713
- [Background] Holmich P. Long-standing groin pain in sportspeople falls into three primary patterns, a "clinical entity" approach: a prospective study of 207 patients. Br J Sports Med. 2007 Apr;41(4):247-52; discussion 252. doi: 10.1136/bjsm.2006.033373. Epub 2007 Jan 29. PMID 17261557
- [Background] Tyler TF, Nicholas SJ, Campbell RJ, McHugh MP. The association of hip strength and flexibility with the incidence of adductor muscle strains in professional ice hockey players. Am J Sports Med. 2001 Mar-Apr;29(2):124-8. doi: 10.1177/03635465010290020301. PMID 11292035
- [Background] Whittaker JL, Small C, Maffey L, Emery CA. Risk factors for groin injury in sport: an updated systematic review. Br J Sports Med. 2015 Jun;49(12):803-9. doi: 10.1136/bjsports-2014-094287. Epub 2015 Apr 1. PMID 25833903
- [Background] Machotka Z, Kumar S, Perraton LG. A systematic review of the literature on the effectiveness of exercise therapy for groin pain in athletes. Sports Med Arthrosc Rehabil Ther Technol. 2009 Mar 31;1(1):5. doi: 10.1186/1758-2555-1-5. PMID 19331695
- [Background] Yousefzadeh A, Shadmehr A, Olyaei GR, Naseri N, Khazaeipour Z. Effect of Holmich protocol exercise therapy on long-standing adductor-related groin pain in athletes: an objective evaluation. BMJ Open Sport Exerc Med. 2018 Jun 26;4(1):e000343. doi: 10.1136/bmjsem-2018-000343. eCollection 2018. PMID 30018787
- [Background] Serner A, van Eijck CH, Beumer BR, Holmich P, Weir A, de Vos RJ. Study quality on groin injury management remains low: a systematic review on treatment of groin pain in athletes. Br J Sports Med. 2015 Jun;49(12):813. doi: 10.1136/bjsports-2014-094256. Epub 2015 Jan 29. PMID 25633830
- [Background] Kalichman L, Ben David C. Effect of self-myofascial release on myofascial pain, muscle flexibility, and strength: A narrative review. J Bodyw Mov Ther. 2017 Apr;21(2):446-451. doi: 10.1016/j.jbmt.2016.11.006. Epub 2016 Nov 14. PMID 28532889
- [Background] Dines JS, Bedi A, Williams PN, Dodson CC, Ellenbecker TS, Altchek DW, Windler G, Dines DM. Tennis injuries: epidemiology, pathophysiology, and treatment. J Am Acad Orthop Surg. 2015 Mar;23(3):181-9. doi: 10.5435/JAAOS-D-13-00148. Epub 2015 Feb 9. PMID 25667400
- [Background] Mauntel TC, Clark MA, Padua DA. Effectiveness of Myofascial Release Therapies on Physical Performance Measurements: A Systematic Review . Athl Train Sport Heal Care. 2014 Jul 1;6(4):189-96.
- [Background] Barnes MF. Efficacy study of the effect of a myofascial release treatment technique on obtaining pelvic symmetry. J Bodyw Mov Ther. 1997 Oct;1(5):289-96.